CLINICAL TRIAL: NCT05107440
Title: BREATHE: A Mixed-methods Evaluation of a Virtual Self-management Program for People Living With Long COVID-19 in Alberta
Brief Title: BREATHE: Virtual Self-management for Long COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: REB21-1359
Record Dates: First submitted 2021-10-13; First posted 2021-11-04 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-01

CONDITIONS: COVID-19
Keywords: Long COVID; Post COVID-19 condition; Post-acute COVID-19 syndrome
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome | interventions — Beclomethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BREATHE (Experimental): This is an eight-week intervention involving two sessions per week, hosted virtually on Zoom. The main session is scheduled to last 60 min and the session hosts remain online for an additional 15 minutes to answer individual questions on the management of symptoms and activities that have not been addressed during the main session. The content was developed based on clinical experience, best available evidence for the management of specific symptoms (chronic fatigue, post-exertional malaise, breathing discomfort) in other conditions, including post-viral syndromes, and the current understanding and recommendations for rehabilitation of people living with long COVID. Long COVID can be isolating, and challenges often interfere with everyday lifestyle and socialization. The investigators have incorporated breakout rooms (where the group is divided into two smaller groups based on current activity limitations) to include elements of peer support.
  Interventions: Other: BREATHE

INTERVENTIONS:
Other: BREATHE — A virtual, multidisciplinary, patient-centred self-management program for long COVID. The BREATHE program provides education on Breathing, Rest/recovery, Education, Activity management, Thinking/cognition, Healthy voice strategies, and Eating/nutrition.

SUMMARY:
A mixed-methods evaluation of a virtual self-management program for people living with long COVID in Alberta.

DETAILED DESCRIPTION:
Background & Rationale

The possible volume of current and future long COVID patients in Alberta is so high (based on the above numbers, more than 20,000) that primary care may not be able to cope given current resources (for example, the waitlist for post-COVID-19 clinics is >3 months). While a Rehabilitation Advice Line and online resources have been created for Albertans with long COVID, many patients are struggling and need more support for self-management to promote recovery. Alongside shortness of breath, long COVID is often characterized by chronic fatigue that is clinically relevant and is at least as severe as fatigue in several other clinical conditions. Other symptoms can include dry cough, cognitive impairment ("brain fog"), heart palpitations, chest tightness, and dizziness. Individuals living with long COVID describe an unpredictable and episodic trajectory with a relapse-remitting nature. Since February 2021, the investigators have been delivering a free virtual program for people with long COVID in Alberta due to an overwhelming demand for physical therapy/support for chronic symptoms. This program has undergone iterative improvements based on new understanding and participant feedback. The program is feasible given the ongoing demand (rapid recruitment of 16-18 participants in three previous programs) and high attendance (>80%). In the most recent cohort, of the participants that responded, 100% found the program helpful, 91% felt more confident about managing symptoms, 91% would recommend the program to other people with long COVID (feedback collected using a brief anonymous survey as part of quality improvement). The objective of this exploratory study is to collect quantitative and qualitative data to evaluate the safety and acceptability of a virtual self-management program for people living with long COVID. Pre-to-post intervention patient-reported outcomes (PROs) will also be collected, and the proportion of participants improving or deteriorating will be reported.

Methods

This is a mixed-methods evaluation of a free, virtual, multidisciplinary, patient-centred self-management program for long COVID. The BREATHE program provides education on Breathing, Rest/recovery, Education, Activity management, Thinking/cognition, Healthy voice strategies, and Eating/nutrition. Two previous pilot iterations of the program took place earlier in 2021, and the BREATHE program in its current format is currently taking place (Aug-Oct, 2021) and will be repeated from Oct-Dec 2021. There is no required in-person element to this study; assessments and program sessions take place virtually via REDCap (secure data collection platform) and Zoom (secure video platform). Participant eligibility criteria were based on the World Health Organization's clinical case definition for post COVID-19 condition.

BREATHE is an eight-week intervention involving two sessions per week, hosted virtually on Zoom. The content was developed based on clinical experience, best available evidence for the management of specific symptoms (chronic fatigue, post-exertional malaise, breathing discomfort, sleep disruption) in other conditions, including post-viral syndromes, and the current understanding and recommendations for rehabilitation of people living with long COVID. The remaining sessions were developed and delivered by content experts (occupational therapist, nutritional consultant, mental health professional) who are familiar with the unique difficulties that people with long COVID face. The investigators have incorporated breakout rooms to include elements of peer support (affirmation of feelings and behaviours, expressions of empathy and reassurance, support for coping with negative emotions, encouraging persistence and optimism). Intervention attendance and adverse events will be reported. Because this is a self-management intervention, the main pre-post outcome of interest is participants' confidence in managing their symptoms and daily activities. Additional outcomes are fatigue, breathing discomfort, functional status and health-related quality of life. To gain participant perspectives on the BREATHE program, participants will be asked to take part in a one-on-one interview via Zoom within two weeks following the final intervention session. A semi-structured interview guide was developed, informed by the Theoretical Framework of Acceptability.

ELIGIBILITY:
Eligibility criteria were based on the World Health Organization's clinical case definition for post-COVID-19 condition, which "occurs in individuals with a history of probable or confirmed Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection, usually 3 months from the onset of COVID-19 with symptoms that last for at least 2 months and cannot be explained by an alternative diagnosis. Common symptoms include fatigue, shortness of breath, cognitive dysfunction but also others which generally have an impact on everyday functioning. Symptoms may be new onset, following initial recovery from an acute COVID-19 episode, or persist from the initial illness. Symptoms may also fluctuate or relapse over time".

Inclusion Criteria:

* Participant has English language fluency (approximately grade 8-10 reading level) and is able to provide informed consent.
* Participant is a resident in Alberta, Canada.
* Participant had confirmed COVID-19 via a positive molecular or antigen test within the past 18 months. Alternatively, in the case of a lack of access to testing, evidence of infection including close contact with a confirmed case of COVID-19 or being linked with a COVID-19 outbreak, or an acute illness including the core symptoms of COVID-19 (cough, fever, shortness of breath, runny nose, sore throat, loss of taste or smell).
* Experiencing symptoms and ongoing functional limitations that have persisted for ≥3 months (from the first positive test/known exposure date/symptom onset). At least one self-reported symptom is fatigue, shortness of breath, cognitive dysfunction or activity intolerance, and
* Post-COVID-19 Functional Status Scale (PFSS) score of ≥2 [22,23].
* Symptoms developed or substantially worsened during or after the acute infection (i.e., they are not explained by a co-occurring condition that pre-dates COVID-19).

Exclusion Criteria:

* Participant does not have access to a smart phone or computer (desktop, laptop, or tablet).
* Receiving ongoing physical therapy via the Workers' Compensation Board.
* Participants are currently participating in a regular rehabilitation program such as the Alberta Health Services (AHS) "Breathe Easy Program - Pulmonary Rehabilitation" or "Supervised Transitional Exercise Program (STEP) Forward - program." Previous participation or being on the waitlist for these services are not exclusion criteria.
* A peripheral oxygen saturation <92% at rest on room air, syncope at rest or on exertion, and any other significant medical complexity that might require medical attention based on clinical judgement.
* A diagnosis of a post-viral syndrome including myalgic encephalomyelitis/chronic fatigue syndrome (ME/CFS) that pre-dates COVID-19.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-10-13 (Actual)

PRIMARY OUTCOMES:
Self-efficacy to manage symptoms | Week 9 i.e. post-intervention (Change from Baseline)
  Total score on the 8-item short form, from the Patient-Reported Outcomes Measurement Information System (PROMIS) Self-efficacy for Managing Chronic Conditions item bank. These PROMIS item banks include all include 8 items that are used to determine a T-score. A T-score of 50 represents the average of people managing chronic health conditions, and ten points is one standard deviation.
Self-efficacy to manage daily activities | Week 9 i.e. post-intervention (Change from Baseline)
  Total score on the 8-item short form, from the PROMIS Self-efficacy for Managing Chronic Conditions item bank
Self-efficacy to manage emotions | Week 9 i.e. post-intervention (Change from Baseline)
  Total score on the 8-item short form, from the PROMIS Self-efficacy for Managing Chronic Conditions item bank

SECONDARY OUTCOMES:
Self-efficacy to manage symptoms | 3-month follow-up (Change from Baseline)
  Total score on the 8-item short form, from the PROMIS Self-efficacy for Managing Chronic Conditions item bank. These PROMIS item banks include all include 8 items that are used to determine a T-score. A T-score of 50 represents the average of people managing chronic health conditions, and ten points is one standard deviation.
Self-efficacy to manage daily activities | 3-month follow-up (Change from Baseline)
  Total score on the 8-item short form, from the PROMIS Self-efficacy for Managing Chronic Conditions item bank
Self-efficacy to manage emotions | 3-month follow-up (Change from Baseline)
  Total score on the 8-item short form, from the PROMIS Self-efficacy for Managing Chronic Conditions item bank
Fatigue severity (FACIT-F) | Week 9 i.e. post-intervention (Change from Baseline)
  Total score on the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Scale
Fatigue severity (FACIT-F) | 3-month follow-up (Change from Baseline)
  Total score on the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Scale
Medical Research Council (MRC) breathlessness scale grade | Week 9 i.e. post-intervention (Change from Baseline)
  Modified according to recommendations for core outcomes for COVID-19 research.
Medical Research Council (MRC) breathlessness scale grade | 3-month follow-up (Change from Baseline)
  Modified according to recommendations for core outcomes for COVID-19 research.
Post-COVID-19 Functional Scale (PCFS) grade | Week 9 i.e. post-intervention (Change from Baseline)
  Post-COVID-19 Functional Scale (PCFS)
Post-COVID-19 Functional Scale (PCFS) grade | 3-month follow-up (Change from Baseline)
  Post-COVID-19 Functional Scale (PCFS)
Recovery grade | Week 9 i.e. post-intervention (Change from Baseline)
  Recommended core outcome measure
Recovery grade | 3-month follow-up (Change from Baseline)
  Recommended core outcome measure
Physical functioning subscale score | Week 9 i.e. post-intervention (Change from Baseline)
  36-Item Short-Form Health Survey
Physical functioning subscale score | 3-month follow-up (Change from Baseline)
  36-Item Short-Form Health Survey
Role limitations due to physical health subscale score | Week 9 i.e. post-intervention (Change from Baseline)
  36-Item Short-Form Health Survey
Role limitations due to physical health subscale score | 3-month follow-up (Change from Baseline).
  36-Item Short-Form Health Survey
Role limitations due to emotional problems subscale score | Week 9 i.e. post-intervention (Change from Baseline)
  36-Item Short-Form Health Survey
Role limitations due to emotional problems subscale score | 3-month follow-up (Change from Baseline)
  36-Item Short-Form Health Survey
Emotional well-being subscale score | Week 9 i.e. post-intervention (Change from Baseline)
  36-Item Short-Form Health Survey
Emotional well-being subscale score | 3-month follow-up (Change from Baseline)
  36-Item Short-Form Health Survey
Social functioning subscale score | Week 9 i.e. post-intervention (Change from Baseline)
  36-Item Short-Form Health Survey
Social functioning subscale score | 3-month follow-up (Change from Baseline)
  36-Item Short-Form Health Survey
Energy/fatigue subscale score | Week 9 i.e. post-intervention (Change from Baseline)
  36-Item Short-Form Health Survey
Energy/fatigue subscale score | 3-month follow-up (Change from Baseline)
  36-Item Short-Form Health Survey
Pain subscale score | Week 9 i.e. post-intervention (Change from Baseline)
  36-Item Short-Form Health Survey
Pain subscale score | 3-month follow-up (Change from Baseline)
  36-Item Short-Form Health Survey
General health subscale score | Week 9 i.e. post-intervention (Change from Baseline)
  36-Item Short-Form Health Survey
General health subscale score | 3-month follow-up (Change from Baseline)
  36-Item Short-Form Health Survey
Physical component score | Week 9 i.e. post-intervention (Change from Baseline)
  36-Item Short-Form Health Survey
Physical component score | 3-month follow-up (Change from Baseline)
  36-Item Short-Form Health Survey
Mental component score | Week 9 i.e. post-intervention (Change from Baseline)
  36-Item Short-Form Health Survey
Mental component score | 3-month follow-up (Change from Baseline)
  36-Item Short-Form Health Survey

OTHER OUTCOMES:
Attendance | The 8-week intervention.
  The number of virtual sessions attended expressed as a percentage of those scheduled (16).
Safety (the number and nature of adverse events) | The 8-week intervention.
  Serious adverse events (defined as any untoward medical occurrence that results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, or results in persistent or significant disability/incapacity) will be reported. Participants will be instructed to report adverse events that occur during or outside of intervention sessions. Adverse events will also be described as severe exacerbation in any symptom that results in further disability or further disruption in the ability to conduct normal life functions (beyond existing disability or disruptions due to long COVID).
Tolerability (change in momentary rating of fatigue) | All sessions in the 8-week intervention.
  0-10 numerical rating of fatigue (ROF) scale, measured pre-post each virtual session.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Culos-Reed, PhD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
A de-identified data set will be made available on the Open Science Framework. Participant information will only be presented in aggregate in manuscripts, and direct and indirect identifiers will be removed from the open dataset to ensure participant anonymity.
Supporting Information: Analytic Code
Time Frame: The de-identified data will be posted when the manuscript is uploaded to a scholarly archiving repository.
Access Criteria: Open access to a de-identified dataset.
URL: https://osf.io/ewkzb/